CLINICAL TRIAL: NCT05887154
Title: Minimal Invasive Microwave Ablation in Early Stage breaST cancER, a Feasibility Study
Brief Title: Non Surgical Treatment (Microwave Ablation) of Breast Cancer
Acronym: MASTER
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Monique Dorrius, Principal Investigator, University Medical Center Groningen
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL76030.042.21; 4901216 (Other Grant/Funding Number: UMCG Kankerresearch fonds)
Record Dates: First submitted 2022-12-15; First posted 2023-06-02 (Actual); Last update posted 2023-06-02 (Actual); Status verified 2023-05

CONDITIONS: Breast Cancer Stage I
Keywords: breast cancer; microwave ablation; MRI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Microwave ablation (Other): Each patient will undergo Microwave ablation of breast tumor before the standard clinical care (surgery)
  Interventions: Device: Microwave ablation

INTERVENTIONS:
Device: Microwave ablation — microwave ablation

SUMMARY:
In the Netherlands approximately one out of seven women will develop breast cancer during her life. Most of these breast cancers are early stage, 40% of the women have stage 1. Stage 1 breast cancer means that the cancer is small (size <2cm) and only in the breast tissue or it might be found in lymph nodes close to the breast. The standard treatment for stage 1 breast cancer is breast conserving surgery (BCS), sentinel lymph node procedure (SLNP) and additional radiotherapy. This standard treatment protocol results in a10 years survival rate of 95% for stage 1 disease. However, nowadays there is a discussion whether these early stage breast cancer could be treated less invasively. To reduce the invasiveness of breast cancer treatment, without compromising breast cancer specific survival, minimally invasive ablation procedure of the breast tumor can be an option for small breast lesions.

Patients with a tumor size<2 cm will undergo ultra guided microwave ablation (MWA) with local anesthesia. After a small incision 2-3 millimeters, an MWA electrode is placed at the end of the tumor with ultrasound guidance. The microwaves in MWA create heat around the needle and destroy the cancer cells. There are several advantages of ablation procedures: it is a minimal invasive technique, with a small or absent cutaneous scar and thereby potentially improving patient quality of life. Furthermore, ablative treatment can be done under local anesthesia and/or conscious sedation instead of general anesthesia and in daycare setting, which can reduce treatment cost. A post procedural MRI (after ablation) can determine whether the ablation procedure of the tumor volume is complete. The purpose of this study is to assess whether minimally invasive microwave ablation (MWA) followed by postprocedural MRI scan can be an alternative treatment for breast surgery in early stage breast cancer. Is the quality of life, the cosmetic outcome, fear of breast cancer recurrence, and costs in patient treated with MWA comparable or better compared to patients treated with breast surgery?

ELIGIBILITY:
Inclusion Criteria:

* age should be 18 years and older
* a solid non-lobular invasive breast tumor with a size <2cm based upon ultrasound and MRI measurements
* without mammographic or MRI evidence of extensive disease
* no involved lymph nodes on ultrasound and MRI scan.

Exclusion Criteria:

* more than one breast tumor,
* (lymph node) metastases
* breast implants
* indication for neoadjuvant chemotherapy.
* pacemaker,
* pregnant
* breastfeeding

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
MWA followed by MRI in breast tumors | 1 year
  MWA will be succesfull if less than 20% of the patients has residual disease

SECONDARY OUTCOMES:
Cosmetic outcome | Timepoints 4 days and 2 weeks after MWA and timepoints 4 days, 2 weeks and 2 months after surgery
  Breast Q questionaire
breast cancer recurrence fear | Timepoints 4 days and 2 weeks after MWA and timepoints 4 days, 2 weeks and 2 months after surgery
  Lerman Breast Cancer Worry scal
Quality of life | Timepoints 4 days and 2 weeks after MWA and timepoints 4 days, 2 weeks and 2 months after surgery
  EuroQol 5D5L

IPD SHARING:
Plan to Share IPD: No